CLINICAL TRIAL: NCT03600740
Title: Advancing Pre-operative Targeting for Deep Brain Stimulation in the Globus Pallidus Internus: Functional Segmentation Based on Probabilistic Tractography
Brief Title: Advancing Pre-operative Targeting for Deep Brain Stimulation in the Globus Pallidus Internus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delays in IRB approval and interval start of a competing study
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erik H. Middlebrooks, M.D., Assistant Professor, Radiology and Neurosurgery, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-002176
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Results first posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Deep Brain Stimulation; Diffusion Tensor Imaging
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- GPi DBS (Experimental): Patients selected to undergo GPi DBS placement will be eligible for enrollment in the study. In addition to standard-of-care tests, subjects will undergo an MRI consisting of the proposed novel imaging protocol prior to placement of DBS. The patient will subsequently undergo standard-of-care therapy for DBS placement. Once the stimulator has been programmed post-operatively, the stimulation parameters and corresponding clinical changes will be collected and used to model the volume of activated tissue. The patient will additionally undergo a follow-up MRI used to localize the electrode within the brain to further localize the volume of activated tissue.
  Interventions: Device: DBS Programming

INTERVENTIONS:
Device: DBS Programming — DBS Programming may be temporarily altered based on imaging data to measure a change in clinical symptoms.

SUMMARY:
In the proposed pilot project, MRI data will be prospectively collected to show the feasibility of the segmentation algorithm and the potential relation to final lead positioning. Patients will be selected from those undergoing GPi DBS placement. This pilot data will serve as a basis for pursuing funding for a larger trial evaluating the prospective ability of the 3T targeting study to improve outcomes and decrease complications in GPi DBS placement. Improved outcomes and patient experience would be expected to further contribute to our facility as a center of excellence for treatment of movement disorders.

ELIGIBILITY:
Patient with the diagnosis of Parkinson's Disease selected for placement of globus pallidus internus (GPi) deep brain stimulator (DBS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik H Middlebrooks, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GPi DBS
Started | 1
Completed | 0
Not Completed | 1
Not completed — Surgical plan was altered-subject not eligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | GPi DBS
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Unified Parkinson's Disease Rating Scale III (UPDRS-III)
Description: Pre-operative and post-operative UPDRS-III will be assessed to measure symptom improvement and correlated with imaging data.
Time Frame: 3 months
Population: Study was terminated due to delays in IRB approval and interval start of a competing study. Surgical plan was altered-subject not eligible. Data was not collected or analyzed.
Arm/Group | GPi DBS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 1 week
Arm/Group | GPi DBS
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Study was terminated due to delays in IRB approval and interval start of a competing study. Surgical plan was altered-subject not eligible. Data was not collected or analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT03600740/Prot_SAP_000.pdf